CLINICAL TRIAL: NCT05403515
Title: Effects of Aromatherapy and Foot Massage on Happiness, Sleep Quality, and Fatigue Levels of Patients With Stroke
Brief Title: Aromatherapy and Foot Massage on Happiness, Sleep Quality, and Fatigue Levels of Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Kevser Sevgi Ünal Aslan, assistant professor, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Osmaniye Korkut Ata Unıvesity
Record Dates: First submitted 2022-05-23; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Stroke, Ischemic
Keywords: Foot massage; Aromatherapy massage; Happiness; Sleep quality; Fatigue
MeSH Terms: conditions — Ischemic Stroke; Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Routine nursing interventions were performed on the patients.
- Foot massage group: (Experimental): For the patients in this group, sociodemographic form, happiness questionnaire, and PSQI was applied as pretest in preliminary examination. The final examination was performed 1 month later (posttest) by using the same scale. For the patients in foot massage group, 30-min foot massage sessions (15 min for each foot, 3 sessions per week for 1 month) were performed in a special room of rehabilitation center, in a quiet atmosphere at suitable temperature and without environmental stimulants.
  Interventions: Other: foot massage
- Foot massage +Aromatherapy group: (Experimental): For the patients in this group, sociodemographic form, happiness questionnaire, and PSQI was applied as pretest in preliminary examination. The final examination was performed 1 month later (posttest) by using the same scale. During the foot massage + aromatherapy lavender inhalation intervention, the patients were given lavender oil for 30 minutes by using a censer. The intervention protocol was developed reviewing the literature about lavender oil inhalation
  Interventions: Other: Foot massage +Aromatherapy group

INTERVENTIONS:
Other: foot massage — foot massage
  Arms: Foot massage group:
Other: Foot massage +Aromatherapy group — foot massage and lavender oil inhalation
  Arms: Foot massage +Aromatherapy group:

SUMMARY:
Background: Stroke puts important economic and social loads on the society and was reported to be the most important reason for disability throughout the world.

Purpose: The present study aims to experimentally examine the effect of aromatherapy and foot massage on happiness, sleep quality, and fatigue levels of patients with stroke.

Material and method: The present study is a randomized clinical study with a control group. Participants were randomly divided into three groups (foot massage + aromatherapy, aromatherapy, and control). The study was carried out with 91 patients diagnosed with stroke. The data were collected using Sociodemographic Status Survey, Oxford Happiness Questionnaire, Piper Fatigue Scale, Pittsburgh Sleep Quality Index (PSQI). Statistical analyses were performed using SPSS (IBM SPSS Statistics 24) package program. The results were interpreted using frequency tables and descriptive statistics. Foot massage group was given 30min foot massage sessions (3 days per week) for 4 weeks, whereas foot massage + aromatherapy group was given lavender oil inhaler during the foot massage.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were diagnosis of stroke at least 3 months, stroke levels of mild or moderate, no use of sleeping pill, volunteering in participation, not being allergic to aromatic oils, no problem with sense of smell, and no lung problem

Exclusion Criteria:

* Exclusion criteria were ulceration or lesion problem in foot, bone deformation in foot, history of allergy, cognitive or mental or language problems, difficulty in verbal communication, psychotic disorders, and not knowing the Turkish language.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
foot massage changes improves happiness and sleep quality. | 1 month
  Oxford Happiness Questionnaire - Short Form (OHQ - S) The total score ranges between 7 and 35 points.
  Pittsburgh Sleep Quality Index (PSQI):
  To identify the sleep is good or bad, PSQI quantitatively measures the quality of sleep. It includes a total of 24 items. Total score of 0-4 points indicates a good sleep quality and the scores between 5 and 21 indicate a poor sleep quality Piper Fatigue Scale Developed by Piper et al. (1998), this scale consists of 24 items and assesses 4 subjective dimensions of fatigue. Reliability and validity of Piper Fatigue Scale for Turkish society were tested by Can (2001). The mean score of 0 point indicates that there was no fatigue, whereas mean scores between 1 and 3 indicate a mild level of fatigue, those between 4 and 6 indicate a moderate level of fatigue, and those between 7 and 10 indicate a severe level of fatigue

SECONDARY OUTCOMES:
Lavender oil inhalation changes happiness and sleep quality | 1 month
  Oxford Happiness Questionnaire - Short Form (OHQ - S) The total score ranges between 7 and 35 points.
  Pittsburgh Sleep Quality Index (PSQI):
  To identify the sleep is good or bad, PSQI quantitatively measures the quality of sleep. It includes a total of 24 items. Total score of 0-4 points indicates a good sleep quality and the scores between 5 and 21 indicate a poor sleep quality Piper Fatigue Scale Developed by Piper et al. (1998), this scale consists of 24 items and assesses 4 subjective dimensions of fatigue. Reliability and validity of Piper Fatigue Scale for Turkish society were tested by Can (2001). The mean score of 0 point indicates that there was no fatigue, whereas mean scores between 1 and 3 indicate a mild level of fatigue, those between 4 and 6 indicate a moderate level of fatigue, and those between 7 and 10 indicate a severe level of fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Sevgi Ü ASLAN, Principal Investigator — OSMANİYE KORKUT ATA UNİVERSİTY
Locations (1):
- Sercan Altın, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data can be shared if the author gives consent for appropriate reasons.